CLINICAL TRIAL: NCT00192179
Title: A Phase II, Prospective, Randomized, Double-Blind, Placebo, Controlled Trial, to Assess the Safety and Tolerability of Influenza Virus Vaccine, Trivalent, Types A & B Live Cold-Adapted Liquid Formulation (CAIV-T) in Healthy Children and Adolescents Ages 6 to Less Than 18 Years.
Brief Title: A Phase II, Trial to Assess the Safety and Tolerability of Influenza Virus Vaccine, CAIV-T in Healthy Children and Adolescents Ages 6 to Less Than 18 Years.
Acronym: FluMist
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Raburn Mallory, MD/ Sr Dir Clinical Development, MedImmune
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D153-P526
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-02

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CAIV-T (Experimental): The total volume of 0.2 ml was administered intranasally with a spray applicator (approximately 0.1 mL into each nostril).
  Interventions: Biological: Cold-adapted influenza vaccine trivalent (CAIV-T)
- Placebo (Placebo Comparator): The total volume of 0.2 ml was administered intranasally with a spray applicator (approximately 0.1 mL into each nostril).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Cold-adapted influenza vaccine trivalent (CAIV-T) — The total volume of 0.2 ml was administered intranasally with a spray applicator (approximately 0.1 ml into each nostril). Each dose of CAIV-T used in this study contained approximately 10^7+/-0.5 fluorescent focus units (FFU) (equivalent to 10^7+/-0.5 TCID50) of each of the following three influenza virus strains: Influenza Cold Adapted Virus Type H1N1, strain A/New Caledonia/20/99; Influenza Cold Adapted Virus Type H3N2, strain A/ Panama/2007/99; Influenza Cold Adapted Virus Type B, strain B/Hong Kong/ 330/01.
  Arms: CAIV-T
Biological: Placebo — The placebo consisted of physiologic normal saline.
  Arms: Placebo

SUMMARY:
A safety study to compare, over a 7 day period, the fever rates following one dose of either Influenza Virus Vaccine or placebo administered outside the influenza season to healthy children and adolescents aged 6 to less than 18 years.

DETAILED DESCRIPTION:
This was a prospective, randomized, double-blind, placebo-controlled, study. Subjects were randomized to receive either CAIV-T or Placebo. All subjects were healthy children and adolescents aged at least 6 years of age and less than 18 years of age at the time of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* who are aged 6 to less than 18 years at the time of enrolment
* who, if female and is of child bearing potential is using reliable method of hormonal and/or non-hormonal contraception (which includes cervical cap, diaphragm, condoms, with spermicide or IUD) during sexual intercourse throughout the entire study period; has provided a negative pregnancy test (with detection limit of less than or equal to 25mL/ml) no more than 24 hours prior to the study vaccine administration and agreed to avoid pregnancy during participation in the study.

N.B.lactating females are excluded from the study.

* who are in good health as determined by medical history, physical examination and clinical judgement
* whose parent(s)/legal guardian(s) have provided written informed consent after the nature of the study has been explained
* who, along with their parent(s)/legal guardian(s) will be available until completion of the study
* whose parent(s)/legal guardian(s), can be reached by study staff for the post vaccination contacts(telephone, clinic or home visit)

Exclusion Criteria:

* who along with their parent(s)/legal guardian(s) are perceived to be unavailable or difficult to contact for evaluation or study visits during the study period
* with any serious chronic disease (e.g. with signs of cardiac or renal failure or severe malnutrition) including progressive neurological disease
* with Down's syndrome or other known cytogenetic disorders
* with a known or suspected disease of the immune system or those receiving immunosuppressive therapy, including systemic corticosteroids; or cytotoxic agents
* who received any blood products, including immunoglobulin, in the period from six months prior to vaccination through to the conclusion of the study
* have an immunosuppressed or an immunocompromised individual living in the same household
* with a documented history of hypersensitivity to egg or egg protein or any other components of CAIV-T or placebo
* who have a history of Guillain-Barre Syndrome (GBS)
* for whom there is intent to administer any other investigational vaccine or agent from one month prior to enrollment through to the conclusion of the study
* who, in the two weeks prior to entry into the study, received a dose of influenza treatment (commercial or investigational)
* who received aspirin (acetylsalicylic acid) or aspirin-containing products in the two weeks prior to enrollment or for which use is anticipated during the study
* who, at anytime prior to study enrollment, received any influenza vaccine (commercial or investigational)
* with asthma requiring regular medical follow up or hospitalization during the preceding year
* with any medical conditions that in the opinion of the investigator might interfere with interpretation of the study results
* Note: Pregnancy in any person who has regular contact with the subjects is not a contraindication to enrollment or ongoing participation of the subject in the study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2003-06; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects with fever greater than or equal to 39.1C oral | Days 0-7

SECONDARY OUTCOMES:
Number of subjects with any reactogenicity | Day 0-7
  Following vaccination the following reactions were reported daily: runny nose/nasal congestion, sore throat, cough, vomiting, decreased activity level, decreased appetite, irritability, abdominal pain together with oral temperature were referred to as prompted systemic reactions.
Number of subjects with any adverse events | Days 0-7
  Adverse events were defined as any untoward, undesired or unexpected clinical event in the form of signs, symptoms, disease or laboratory or physiological observations that occurred in a temporal relationship to the use of a WVR product, regardless of causal relationship.
Number of subjects with any serious adverse events | Days 0-21
  A Serious AE was an AE that occurred after any dose that: resulted in death, regardless of cause; was life-threatening; required in-patient hospitalization or prolonged an existing hospitalization; resulted in a persistent or significant disability or incapacity; resulted in cancer; resulted in a congenital anomaly or birth defect (in the offspring of a vaccine recipient, where applicable).

CONTACTS AND LOCATIONS:
Overall Officials: Raburn Mallory, M.D., Study Director — MedImmune LLC
Locations (6):
- Belgium (3):
  - Catholic University Leuven, Leuven
  - Zamenhoflaan 12, Schoten
  - Universiteit Antwerpen, Wilrijk
- Oddzial Dzieciecy Szpitala Powiatowete im, Trzebnica, Poland
- United Kingdom (2):
  - The Gables Medicentre, Coventry
  - Townhead Surgery, Irvine, Ayshire